CLINICAL TRIAL: NCT07120438
Title: Comparison Between Diaphragmatic Ultrasound and Rapid Shallow Breathing Index (RSBI) in Predicting Weaning Success in Patients on Mechanical Ventilation for More Than 48 Hours in the ICU of Dr. Sardjito Hospital, Yogyakarta
Brief Title: Comparison of Diaphragm Ultrasound and RSBI for Predicting Weaning Success in Mechanically Ventilated ICU Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Meta Restu Synthana, Fellow in Intensive Care, Gadjah Mada University
Other Study IDs: METAKIC
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ventilator Weaning; Mechanical Ventilation; Respiratory Insufficiency Requiring Mechanical Ventilation; Weaning From Mechanical Ventilation; Weaning From Mechanical Ventilation in Care Unit; Intensive Care Unit Patients
Keywords: Diaphragmatic Ultrasound; Rapid Shallow Breathing Index; Diaphragm Thickening Fraction; Diaphragm Excursion; Weaning Prediction; ICU; Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Patients on Mechanical Ventilation >48 Hours: This cohort includes adult patients admitted to the Intensive Care Unit (ICU) who have been on mechanical ventilation for more than 48 hours. Each participant undergoes assessment using both the Rapid Shallow Breathing Index (RSBI) and diaphragm ultrasonography, including measurements of diaphragmatic excursion (DE) and diaphragmatic thickening fraction (DTF). These assessments are conducted prior to extubation to evaluate their predictive accuracy in determining weaning success or failure.

SUMMARY:
The goal of this observational study is to evaluate the predictive value of diaphragmatic ultrasound compared to the Rapid Shallow Breathing Index (RSBI) in determining weaning success among mechanically ventilated patients in the ICU for more than 48 hours.

The main question it aims to answer is:

Which is more effective in predicting weaning success: diaphragmatic ultrasound (including Diaphragmatic Excursion [DE] and Diaphragm Thickening Fraction [DTF]) or RSBI, in patients ventilated >48 hours in the ICU of Dr. Sardjito General Hospital, Yogyakarta?

Participants will be adult ICU patients who are undergoing weaning from mechanical ventilation after more than 48 hours. Before extubation, each participant will undergo diaphragmatic ultrasound assessment to measure DE and DTF, along with RSBI measurement. The predictive accuracy of these parameters will be evaluated by comparing them with the actual weaning outcomes.

Secondary objectives include:

1. Assessing whether diaphragmatic ultrasound is associated with a higher weaning success rate than RSBI.
2. Evaluating the correlation between DE values and successful weaning.
3. Determining the optimal cutoff values of DE and DTF as predictors of weaning failure.
4. Analyzing the incidence of weaning failure in patients who do not meet optimal diaphragm function criteria.
5. Identifying DE and DTF thresholds that may help reduce the risk of reintubation.

DETAILED DESCRIPTION:
This observational cohort study aims to investigate the diagnostic utility of diaphragm ultrasound (specifically diaphragmatic excursion (DE) and diaphragm thickening fraction (DTF)) as alternative weaning predictors in adult ICU patients undergoing mechanical ventilation for more than 48 hours. Given the limitations of the Rapid Shallow Breathing Index (RSBI) in predicting weaning outcomes, ultrasound-based parameters offer a promising physiological assessment tool by directly evaluating diaphragmatic function.

Diaphragm ultrasound will be performed within a defined period prior to planned weaning, following standardized imaging protocols to obtain DE and DTF measurements. All ultrasound assessments will be conducted by trained clinicians using point-of-care ultrasound devices available in the ICU. These values will be compared with the corresponding RSBI obtained as part of routine care, without interfering with the clinical decision-making process.

The study will analyze predictive accuracy metrics (such as sensitivity, specificity, and area under the receiver operating characteristic curve) to compare RSBI with diaphragm ultrasound indices. Subgroup analyses will assess the relationship between suboptimal diaphragm function and weaning failure, as well as evaluate threshold values of DE and DTF that may serve as reliable predictors for extubation outcomes. The study will also explore how these indices correlate with rates of reintubation and prolonged weaning.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been on mechanical ventilation for more than 48 hours
2. Adult patients aged ≥18 years
3. Patients who meet the criteria for hemodynamic stability for weaning
4. Patients or their families have provided written informed consent
5. Patients with FiO₂ < 50%, PEEP level < 5 cm H₂O, respiratory rate < 30 breaths per minute, PaO₂/FiO₂ > 200, and GCS > 13
6. Patients who have successfully completed the Spontaneous Awakening Trial (SAT) and Spontaneous Breathing Trial (SBT)

Exclusion Criteria:

1. Patients with neuromuscular disorders, anatomical abnormalities of the diaphragm, or diaphragmatic palsy
2. Patients with a history of severe thoracic trauma affecting diaphragm function on one or both sides
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects who meet the predetermined criteria. The target population refers to the broader group to which the results of this study are intended to be applied. This population is general in nature but limited by clinical and demographic characteristics. The accessible population is a subset of the target population, defined by place and time, which can be reached by the researcher and will ultimately serve as the source of study participants (Sastroasmoro and Ismail, 2008).The target population in this study comprises adult male and female patients who are on mechanical ventilation in the Intensive Care Unit (ICU) at Dr. Sardjito Hospital, Yogyakarta. The accessible population includes patients with indications for weaning from mechanical ventilation in the ICU of Dr. Sardjito Hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Extubation Success Rate | After extubation
  Proportion of patients who remain extubated for at least 48 hours following planned extubation.

SECONDARY OUTCOMES:
Diagnostic Accuracy of RSBI, Diaphragmatic Excursion, and Diaphragmatic Thickening Fraction (DTF) for Predicting Extubation Success | Prior to extubation
  Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) will be calculated for diaphragmatic excursion and diaphragmatic thickening fraction (ΔTdi%) to predict successful weaning from mechanical ventilation. Receiver Operating Characteristic (ROC) curve analysis will be used to evaluate and compare the clinical utility of RSBI, diaphragmatic excursion, and DTF in predicting extubation success.

IPD SHARING:
Plan to Share IPD: Undecided